CLINICAL TRIAL: NCT03216499
Title: Single-Arm, Open-Label Phase II Efficacy Study of First-in-Class HIF-2 Alpha Inhibitor, PT2385, for Patients With Recurrent Glioblastoma
Brief Title: HIF-2 Alpha Inhibitor PT2385 in Treating Patients With Recurrent Glioblastoma
Acronym: PT2385
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Peloton Therapeutics, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABTC 1602; IRB00132128 (Other: JHM IRB); UM1CA137443 (NIH)
Record Dates: First submitted 2017-07-11; First posted 2017-07-13 (Actual); Results first posted 2020-09-21 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-01

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — PT2385; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (HIF-2 alpha inhibitor PT2385) (Experimental): Patients receive HIF-2 alpha inhibitor PT2385 PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Pharmacological Study
  Laboratory Biomarker Analysis
  Pharmacogenomic Study
  Interventions: Drug: HIF-2alpha Inhibitor PT2385; Other: Pharmacological Study; Other: Laboratory Biomarker Analysis; Other: Pharmacogenomic Study

INTERVENTIONS:
Drug: HIF-2alpha Inhibitor PT2385 — Given PO
  Other Names: HIF-2alpha Inhibitor PT2385, PT2385
Other: Pharmacological Study — Correlative studies
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacogenomic Study — Correlative studies
  Other Names: PHARMACOGENOMIC, Pharmacogenomic Study

SUMMARY:
This phase II trial studies how well HIF-2 alpha inhibitor PT2385 works in treating patients with recurrent glioblastoma. HIF-2 alpha inhibitor PT2385 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the efficacy of hypoxia inducible factor (HIF)-2 alpha inhibitor PT2385 (PT2385) as measured by radiographic response rate (by Response Assessment in Neuro-Oncology, RANO, criteria) in patients with recurrent glioblastoma.

SECONDARY OBJECTIVES:

I. To estimate the efficacy of PT2385 as measured by progression free and overall survival in patients with recurrent glioblastoma.

II. To determine the safety of oral PT2385 in patients with recurrent glioblastoma.

TERTIARY OBJECTIVES:

I. To describe the pharmacokinetic and pharmacodynamic properties of PT2385 in patients with recurrent glioblastoma.

II. To describe baseline intratumoral hypoxia using novel, advanced magnetic resonance (MR)-based neuroimaging sequences in patients with recurrent glioblastoma.

III. To explore genetic polymorphisms involved in the metabolism of PT2385.

OUTLINE:

Patients receive HIF-2 alpha inhibitor PT2385 orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months for 2 years and every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* • Patients must have histologically confirmed glioblastoma that is progressive or recurrent following radiation therapy and temozolomide according to the Response Assessment in Neuro-Oncology (RANO) criteria with:

  * New contrast-enhancing lesion outside of radiation field on decreasing, stable, or increasing doses of corticosteroids
  * Increase by >= 25% in the sum of the products of perpendicular diameters between the postradiotherapy scan with the smallest tumor measurement and a scan at least 12 weeks from completion of radiation therapy (RT) + temozolomide (TMZ), on stable or increasing doses of corticosteroids

    ** Note: clinical deterioration not attributable to concurrent medication or comorbid conditions is sufficient to declare progression on current treatment but not for entry onto a clinical trial for recurrence
    * Tumor O(6)-methylguanine-DNA-methyltransferase (MGMT) methylation status must be available; results of routinely used methods for MGMT methylation testing (e.g. mutagenically separated polymerase chain reaction, (MSPCR), or quantitative polymerase chain reaction (PCR)) are acceptable
    * Patients must have a tumor tissue form indicating availability of archived tissue from a previous surgery for glioblastoma, completed and signed by a pathologist
    * Patients must have measurable (defined by at least 1 cm x 1 cm) contrast-enhancing disease by magnetic resonance imaging (MRI) imaging within 21 days of starting treatment
    * Patients must be able to undergo MRI of the brain with gadolinium; patients must be maintained on a stable or decreasing dose of corticosteroid regimen (no increase for 5 days) prior to this baseline MRI
    * Patients must be in first recurrence of glioblastoma following radiation therapy and temozolomide
    * Patients must have recovered from severe toxicity of prior therapy; the following intervals from previous treatments are required to be eligible:
  * 12 weeks from the completion of radiation
  * 6 weeks from a nitrosourea chemotherapy
  * 3 weeks from a non-nitrosourea chemotherapy
  * 4 weeks from any investigational (not Food and Drug Administration (FDA)-approved) agents
  * 2 weeks from administration of a non-cytotoxic, FDA-approved agent (e.g., erlotinib, hydroxychloroquine, etc.)

    * Patients must have a Karnofsky performance status >= 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
    * Absolute neutrophil count >= 1,500/microliter (mcL)
    * Platelets >= 100,000/mcL
    * Hemoglobin >= 9 g/dL
    * Total bilirubin =< institutional upper limit of normal
    * Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase (SGOT))/ alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase (SGPT)) =< 4 x institutional upper limit of normal
    * Creatinine =< institutional upper limit of normal OR creatinine clearance >= 60 ml/min/1.73m^2 for patients with creatinine levels above institutional normal
    * Activated partial thromboplastin time (APTT) or partial thromboplastin time (PTT) =< 1.5 x institutional upper limit of normal
    * Patients must be able to provide written informed consent
    * Women of childbearing potential must have a negative serum pregnancy test prior to study start; women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and through 30 days after the last dose of study drug; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and through 30 days after the last dose of study drug
    * Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder; patients with prior malignancies must be disease-free for >= five years
    * Patients must be able to swallow tablets

Exclusion Criteria:

* • Patients receiving any other investigational agents are ineligible

  * Patients must not have received prior anti- Vascular endothelial growth factor (VEGF) therapy including bevacizumab (i.e. patients must be bevacizumab naive)
  * Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to PT2385 are ineligible
  * Patients on enzyme-inducing anti-epileptic drugs (EIAED) are not eligible for treatment on this protocol; patients may be on non-enzyme inducing anti-epileptic drugs or not be taking any anti-epileptic drugs; patients previously treated with EIAED may be enrolled if they have been off the EIAED for 10 days or more prior to the first dose of PT2385
  * Patients with a history of bleeding diathesis are ineligible
  * Patients who have not recovered to < Common Terminology Criteria for Adverse Events (CTCAE) grade 2 toxicities related to prior therapy are ineligible
  * Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, clinically significant cardiac disease, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, are ineligible
  * Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with PT2385
  * Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible due to potential drug-drug interactions with PT2385

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Strowd, MD, Study Chair — Wake Forest /ABTC
Locations (10):
- United States (10):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Abrams Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Strowd R, Ellingson B, Raymond C, Yao J, Wen PY, Ahluwalia M, Piotrowski A, Desai A, Clarke JL, Lieberman FS, Desideri S, Nabors LB, Ye X, Grossman S. Activity of a first-in-class oral HIF2-alpha inhibitor, PT2385, in patients with first recurrence of glioblastoma. J Neurooncol. 2023 Oct;165(1):101-112. doi: 10.1007/s11060-023-04456-7. Epub 2023 Oct 21. PMID 37864646

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment Sept 14, 2017 - March 9, 2018, all glioblastoma multiforme (GBM) patients
Groups:
- Treatment (HIF-2 Alpha Inhibitor PT2385): Patients receive hypoxia inducible factor (HIF)-2 alpha inhibitor PT2385 per os (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Pharmacological Study
  Laboratory Biomarker Analysis
  Pharmacogenomic Study
  HIF-2 alpha Inhibitor PT2385: Given PO
  Pharmacological Study: Correlative studies
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacogenomic Study: Correlative studies
Period: Overall Study
Arm/Group | Treatment (HIF-2 Alpha Inhibitor PT2385)
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (HIF-2 Alpha Inhibitor PT2385): Patients receive HIF-2 alpha inhibitor PT2385 PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Pharmacological Study
  Laboratory Biomarker Analysis
  Pharmacogenomic Study
  HIF-2alpha Inhibitor PT2385: Given PO
  Pharmacological Study: Correlative studies
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacogenomic Study: Correlative studies
Arm/Group | Treatment (HIF-2 Alpha Inhibitor PT2385)
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: years] | 62.1 [38.7 to 76.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 1
MGMT Promoter Status [Count of Participants; unit: Participants] — O[6]-methylguanine-DNA methyltransferase (MGMT) is a DNA repair enzyme. In newly diagnosed glioblastomas, the presence of MGMT promoter methylation has been shown to be an independent favorable prognostic factor and a strong predictor of responsiveness to alkylating chemotherapy. The MGMT status reported is either methylated, not methylated or indeterminate.
  Participants
    Methylated | 11
    Not Methylated | 12
    Indeterminate | 1
Extent of tumor resection [Count of Participants; unit: Participants]
  Biopsy | 2
  Subtotal resection | 8
  Gross total resection | 14
Karnofsky Performance Status Score [Median (Full Range); unit: score on a scale] — The Karnofsky Performance Status score is a standard way of measuring the ability of cancer patients to perform ordinary tasks with a score range from 0 to 100. A higher score means patient is better able to carry out daily activities: "100 - Normal; no complaints, no evidence of disease; 90 - Able to carry on normal activity; minor signs or symptoms of disease, 80 - Normal activity with effort; some signs or symptoms of disease; 70 - Cares for self, unable to carry on normal activity or to do active work; 60 - Requires occasional assistance, but is able to care for most of personal needs"
  score on a scale | 80 [70 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Tumor Radiographic Response as Assessed by the RANO Criteria
Description: Tumor radiographic response assessed by Response Assessment in Neuro-Oncology (RANO) criteria.
  * Complete Response (CR) = no change in size of T1-gadolinium-enhancing (T1-Gd+) disease, stable or reduced T2/FLAIR signal, no new lesion, no corticosteroid use, and stable or improved clinical status
  * Partial Response (PR) = ≥50% change in size of T1-Gd+ disease, stable or reduced T2/FLAIR signal, no new lesion, stable or reduced corticosteroid use, and stable or improved clinical status
  * Stable Disease (SD) = <50% reduction to <25% increase size of T1-Gd+ disease, stable or reduced T2/FLAIR signal, no new lesion, stable or reduced corticosteroid use, and stable or improved clinical status
  * Progressive Disease (PD) = ≥25% increase size of T1-Gd+ disease, or increased T2/FLAIR signal, or presence of new lesion, or worsening clinical status.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (HIF-2 Alpha Inhibitor PT2385)
Number analyzed (Participants) | 24
Participants
  complete response | 0
  partial response | 0
  stable | 7
  progression | 17

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS (in months) will be estimated using Kaplan-Meier method along with 95% confidence interval. Definition of PFS is date treatment started to the date of progression.
Time Frame: Assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (HIF-2 Alpha Inhibitor PT2385)
Number analyzed (Participants) | 24
months | 1.8 [1.6 to 2.5]

3. Secondary Outcome: Overall Survival
Description: Overall survival (in months) will be estimated using Kaplan-Meier method along with 95% confidence interval.
Time Frame: From the date of treatment start to the date of death occurrence/or censored at the time of last known alive, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (HIF-2 Alpha Inhibitor PT2385)
Number analyzed (Participants) | 24
months | 7.7 [4.9 to 12.6]

4. Secondary Outcome: Incidence of Grade 3 and Grade 4 Adverse Events
Description: Number of participants experiencing grade 3 and grade 4 adverse events assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (HIF-2 Alpha Inhibitor PT2385)
Number analyzed (Participants) | 24
Participants
  grade 3 anemia | 1
  grade 3 Hyperglycemia | 1
  grade 3 hyponatremia | 2
  grade 3 Hypoxia | 2
  grade 4 Hypoxia | 1

5. Other Pre Specified Outcome: Pharmacokinetics (Cmin) for PT2385
Description: Minimum concentration (Cmin) on Day 15 of cycle 1.
  * Cycle 1, Week 1, Day 1, Pre-dose 1: within 15 minutes prior to dose
  * Cycle 1, Week 1, Day 1, 6 Hours Post-dose 1: 6 hours +/- 15 minutes post-dose
  * Cycle 1, Week 3, Day 15, Pre-dose 1: within 30 minutes prior to dose
Time Frame: Day 15 cycle 1
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Pharmacokinetics for PT2385 Drug Exposure
Description: Drug exposure levels in 3 groups: Cmin >1000ng/mL; Cmin: 300-1000 ng/mL and Cmin <300ng/mL
Time Frame: Day 15 cycle 1
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Determine Association Between Baseline Tumor Acidity and PT2385 (Imaging)
Description: Baseline Tumor acidity was measured using pH-weighted amine chemical exchange saturation transfer (CEST) MRI contrast on the Magnetic Resonance Imaging R^2 = "reversible transverse relaxation rate" (and is proportional to oxygen extraction and thus hypoxia).
  MTR = MTRasym "the asymmetry in the magnetization transfer ratio at 3ppm from water" (and it is a surrogate of tumor acidity (MTR) pH quantitative measure of the acidity or basicity (pH) of aqueous or other liquid solutions. Lower pH values correspond to solutions which are more acidic in nature, while higher values correspond to solutions which are more basic or alkaline.
  Exp = exposure Acid = Acidity Perit Tiss = Peritumoral Tissue Enh Tum = Enhancing Tumor DurTx = Duration treatment
Time Frame: At baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Approximately 1 year
Arm/Group | Treatment (HIF-2 Alpha Inhibitor PT2385)
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 6/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (HIF-2 Alpha Inhibitor PT2385) (N=24)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (HIF-2 Alpha Inhibitor PT2385) (N=24)
aniema (Blood and lymphatic system disorders) | 11 (30)
confusion (Psychiatric disorders) | 4 (4)
Dysphasia (Nervous system disorders) | 2 (2)
Edema Limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 7 (7)
Hyponatremia (Metabolism and nutrition disorders) | 2 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (6)
lymphocyte decrease (Investigations) | 2 (6)
muscle weakness (Nervous system disorders) | 4 (6)
Nausea (Gastrointestinal disorders) | 5 (5)
platelet count decrease (Investigations) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT03216499/Prot_SAP_000.pdf